CLINICAL TRIAL: NCT01417299
Title: The Impact of RPh201 on CVS Patients: Clinical and fMRI Measurements
Acronym: CVS
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This record is an additional copy of the study listed above
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr. Netta Levin, Hadassah Medical Organization, Jerusalem, Israel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0260-11-HMO
Record Dates: First submitted 2011-08-15; First posted 2011-08-16 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2011-08

CONDITIONS: Chronic Vegetative State
Keywords: chronic vegetative state; RPh201; functional MRI
MeSH Terms: conditions — Persistent Vegetative State | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- RPh201 group (Active Comparator): Patients will receive 400 microliter s.c., of RPh201 twice a week for 3 months
  Interventions: Dietary Supplement: RPh201
- placebo group (Placebo Comparator): Patients will receive 400 microliter s.c., of saline twice a week for 3 months
  Interventions: Dietary Supplement: saline

INTERVENTIONS:
Dietary Supplement: RPh201 — Patients will receive 400 microliter s.c., of RPh201 twice a week for 3 months
  Arms: RPh201 group
Dietary Supplement: saline — Patients will receive 400 microliter s.c., of saline twice a week for 3 months
  Arms: placebo group

SUMMARY:
The investigators are studying the impact of RPh201 on chronic vegetative patients. RPh201 has been reported to induce neuronal regeneration in animal models. Evaluation will be done by combining clinical /behavioral assessment with fMRI studies.

ELIGIBILITY:
Inclusion Criteria:

* Chronic vegetative patients

Exclusion Criteria:

* Inability to go through an MRI scans (i.e. metal implants, neurotransmitters)and pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
change in the awareness status of the patients. | 3-6 months
  Clinical and laboratory assessment will be done every two weeks along the treatment period fMRI assessment will be performed 3 times: before the treatment, immediate afterwards and one month following treatment cessation.

SECONDARY OUTCOMES:
change in the awareness status of the patients. | 1 month following the end of the trial
  clinical and fMRI assessment will be performed 1 month following treatment cessation

CONTACTS AND LOCATIONS:
Overall Officials: Tamir Ben-Hur, MD PhD, Principal Investigator — Hadassah Medical Organization